CLINICAL TRIAL: NCT02602860
Title: A Single-center, Open-label Positron Emission Tomography Study to Evaluate the Time-course of Displacement of [11C]UCB-J by Brivaracetam and Levetiracetam in Healthy Volunteers
Brief Title: A Brain Imaging Study With Positron Emission Tomography and the Radiotracer [11C]UCB-J to Estimate How Fast Brivaracetam and Levetiracetam Enter the Brain in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: PRA Health Sciences (Industry); Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EP0074
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
Keywords: SV2A; Levetiracetam; Brivaracetam; PET
MeSH Terms: interventions — 1-((3-(methylpyridin-4-yl)methyl)-4-(3,4,5-trifluorophenyl)pyrrolidin-2-one; brivaracetam; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental): Cohort 1: Half of the subjects will receive LEV as a 5 minute iv infusion during the second Positron Emission Tomography (PET) scan, 60 minutes after the start of [11C]UCB-J administration.
  Cohort 2: Half of the subjects will receive LEV as a 5 minute iv infusion during the first PET scan, 60 minutes after the start of [11C]UCB-J administration. The dose of LEV (500 mg to 2500 mg) or BRV (50 mg to 200 mg) will be decided based on the data obtained in Cohort 1. Subjects will return for a second PET imaging session (Visit 4), 7 to 28 days after completion of their first session (Visit 3) to enter the BRV arm.
  Interventions: Radiation: [11C]UCB-J; Drug: Levetiracetam
- Brivaracetam (Experimental): Cohort 1:Half of the subjects will receive BRV as a 5 minute iv infusion during the second Positron Emission Tomography (PET) scan, 60 minutes after the start of [11C]UCB-J administration.
  Cohort 2:Half of the subjects will receive BRV as a 5 minute iv infusion during the first PET scan, 60 minutes after the start of [11C]UCB-J administration. The dose of BRV (50-200 mg) will be decided based on the data obtained in Cohort 1. Subjects will return for a second PET imaging session,7 to 28 days after completion of their first session to enter the LEV arm.
  Cohort 3:void Cohort 4:Subjects will take oral BRV (25-100 mg bid) for 4 days and a single dose of BRV on Day 5. Pre-/post-block scans will be obtained at the first dose, one post-block scan after the last dose. Additional post-block scans may be obtained 8-10 and 28h or later after last dose; if last scan not needed, subject will return 7 to 28 days later for a post-block scan. Dose range for LEV in Cohort 4 will be 250 to <1500mg.
  Interventions: Radiation: [11C]UCB-J; Drug: Brivaracetam

INTERVENTIONS:
Radiation: [11C]UCB-J — * Pharmaceutical form: Sterile solution for intravenous infusion
  * Concentration: 20 mCi
  * Route of Administration: iv
  Other Names: [11C]APP311
Drug: Brivaracetam — * Pharmaceutical form: Sterile solution for intravenous infusion
  * Concentration: 10 mg/ml
  * Route of Administration: iv
  Other Names: UCB34714
  Arms: Brivaracetam
Drug: Levetiracetam — * Pharmaceutical form: Sterile solution for intravenous infusion
  * Concentration: 100 mg/ml
  * Route of Administration: iv
  Other Names: Keppra; L059
  Arms: Levetiracetam
Drug: Brivaracetam — * Pharmaceutical form: Tablets for oral intake
  * Concentration: 25 mg
  * Route of Administration: oral
  Other Names: UCB34714
  Arms: Brivaracetam

SUMMARY:
This study will estimate how fast two antiepileptic drugs (Levetiracetam and Brivaracetam) enter the human brain. Brain imaging will be used to measure how quickly the radioactive probe [11C]UCB-J exits the brain when Levetiracetam or Brivaracetam are given. This will be used to estimate how fast the antiepileptic drugs enter the brain.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Subject is male or female and between 18 to 55 years of age (inclusive)
* Subject is in good physical and mental health, in the opinion of the Investigator, determined on the basis of medical history, physical and neurological examinations, vital signs, 12-lead Electrocardiography (ECG), and clinical laboratory tests
* Female subjects of childbearing potential must have a negative pregnancy test; female subjects of childbearing potential have to confirm that, for 1 month prior to the first administration of the study medication and during the entire study until the Safety Follow-Up (SFU) Visit she will either use a highly effective contraceptive method (eg, oral contraception, intrauterine device, diaphragm with spermicide) or abstain from sexual activity that can cause pregnancy

Exclusion Criteria:

Exclusion Criteria:

* History or presence of clinically significant respiratory, gastrointestinal, renal, hepatic, pancreatic, hematological, cardiovascular, musculoskeletal, genitourinary, immunological, or dermatological disorders, or any type of cancer
* Subject has a history of a neurological diagnosis, including but not limited to stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, or any other neurological disorder that may influence the outcome or analysis of the scan results
* History of donation of more than 450 mL of blood within 60 days prior to dosing in the Yale PET center or planned donation before 30 days has elapsed since intake of study drug
* The subject has Magnetic Resonance Imaging -incompatible (MRI - incompatible) implants and other contraindications for MRI, such as a pacemaker, artificial joints, non-removable body piercings, etc.
* Subjects who have received a diagnostic or therapeutic radiopharmaceutical less than 7 days prior to participation in this study
* Participation in other recent research studies < 1 month or < 1 year for studies involving ionizing radiation that would cause the subject to exceed the yearly dose limits for healthy volunteers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Level of synaptic vesicle glycoprotein 2A (SV2A) receptor occupancy during the displacement scans | Displacement scans (120 minutes)
  The receptor occupancy will be determined using occupancy plots from the apparent volume of distribution, Vapp values.
Equilibrium tissue to plasma activity ratio (VT) of [11C]UCB-J | Baseline (120 minutes) and Displacement scans (120 minutes)
  The equilibrium tissue to plasma activity ratio (VT) will be used to quantify [11C]UCB-J binding in each brain region of interest before and after administration of Brivaracetam and Levetiracetam.
Tracer displacement halftimes | Baseline (120 minutes) and Displacement scans (120 minutes)
  Tracer displacement halftimes will be estimated from Displacement scans and Baseline scans on the average standardized uptake value (SUV) for all regions over time during 60-minute timeframe.
Tracer-exit corrected halftimes of Brivaracetam or Levetiracetam entry | Baseline (120 minutes) and Displacement scans (120 minutes)
  Tracer-exit corrected halftimes of Brivaracetam or Levetiracetam entry will be estimated by subtracting the tracer clearance halftime from the displacement halftime.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1-844-599-2273(UCB)
Locations (1):
- Ep0074 001, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Finnema SJ, Rossano S, Naganawa M, Henry S, Gao H, Pracitto R, Maguire RP, Mercier J, Kervyn S, Nicolas JM, Klitgaard H, DeBruyn S, Otoul C, Martin P, Muglia P, Matuskey D, Nabulsi NB, Huang Y, Kaminski RM, Hannestad J, Stockis A, Carson RE. A single-center, open-label positron emission tomography study to evaluate brivaracetam and levetiracetam synaptic vesicle glycoprotein 2A binding in healthy volunteers. Epilepsia. 2019 May;60(5):958-967. doi: 10.1111/epi.14701. Epub 2019 Mar 29. PMID 30924924